CLINICAL TRIAL: NCT00478478
Title: Merci Registry - Real World Use of the Merci Retrieval System in Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: INT-REG-001
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemic; Thrombus; Embolectomy; Thrombectomy; Merci; Concentric; Embolus; Embolism; Mechanical
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia; Thrombosis; Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Ischemic Stroke patients: Patients presenting with signs and symptoms consistent with a diagnosis of Acute Ischemic Stroke, who are treated with the Merci Retrieval System during a Mechanical Thrombectomy procedure.
  Interventions: Procedure: Mechanical Thrombectomy

INTERVENTIONS:
Procedure: Mechanical Thrombectomy — Thrombectomy performed with the Merci Retriever in the setting of acute ischemic stroke.
  Other Names: Merci Retrieval System

SUMMARY:
Post-Market Registry on Use of Merci Retrieval System. Primary data to be collected will include:

* Post-procedure revascularization success
* 90-day mRS 0-2
* 90-day mortality

DETAILED DESCRIPTION:
The Merci Registry is a prospective multicenter registry with up to 3000 patients enrolled at a maximum of 100 sites.

The registry requires use (at least one pass in the intracranial vasculature) of any Merci Retriever device (X Series, L Series, V Series) in the setting of acute ischemic stroke due to large vessel intracranial occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient with ischemic stroke is treated with a Merci Retriever that is indicated for thrombus removal in ischemic stroke. "Treated" is defined as being when a Merci Retriever is deployed in the neurovasculature of a patient with an ischemic stroke
* Patient/patient's surrogate provides informed consent and is willing to comply with the protocol requirements and complete required clinical evaluations, or in the absence of informed consent, an IRB/EC approved waiver of consent and executed data use agreement are in place

Exclusion Criteria:

-There are no exclusion criteria for this protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with ischemic stroke treated with a Merci Retriever either alone or in combination with adjunctive therapies such as lytics will be included in the Registry.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2007-06; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Post-procedure revascularization success | post-procedure

SECONDARY OUTCOMES:
NIHSS change from baseline to 24-hours | 24-hour
90-day mRS outcomes | 90-day
90-day mortality | 90-day

CONTACTS AND LOCATIONS:
Overall Officials: Wade S Smith, MD, PhD, Principal Investigator — University of California at San Francisco, SF, CA; Marilyn M Rymer, MD, Principal Investigator — MABSI St. Luke's, Kansas City, MO
Locations (1):
- St. Luke's Brain and Stroke Institute, Kansas City, Missouri, United States

REFERENCES:
- See also: Stryker Neurovascular — http://www.stryker.com/neurovascular